CLINICAL TRIAL: NCT07359911
Title: Effect of A Multimodal Exercise Intervention on Chemotherapy Uptake in Newly Diagnosed Pediatric and AYA Sarcoma Patients (ACTIVE-SARC)
Brief Title: Effect of A Multimodal Exercise Intervention on Chemotherapy Uptake in Newly Diagnosed Pediatric and AYA Sarcoma Patients
Acronym: ACTIVE-SARC
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: Florida Department of Health (Other Government)
Responsible Party: Principal Investigator, Tracy E Crane, PhD, RDN, Associate Professor, University of Miami
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 20250858
Record Dates: First submitted 2026-01-14; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Sarcoma
Keywords: Pediatric; Adolescent; Young Adult
MeSH Terms: conditions — Sarcoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise Intervention Group (EXE) (Experimental): Participants in this group will undergo supervised multimodal (aerobic, resistance, balance) moderate-to-vigorous exercise intervention three 3 times per week for 12 weeks, a total of 36 sessions.
  Total participation duration is about 12 weeks.
  Interventions: Behavioral: Exercise Intervention; Behavioral: Exit Interview
- Usual Care Control Group (UC) (Other): Participants in this group may opt to receive a weekly brief symptom self-assessment as a survey.
  Total participation duration is about 12 weeks.
  Interventions: Behavioral: Usual Care Control

INTERVENTIONS:
Behavioral: Exercise Intervention — Each session will include a brief conversation and standardized symptom assessment, followed by a warm-up including stretching & balance exercises, then a series of resistance exercises, ending with light-moderate intensity aerobic exercise (walking), with a target goal of 45-60 minutes total per session as tolerated by the patient.
  Arms: Exercise Intervention Group (EXE)
Behavioral: Usual Care Control — A weekly brief symptom self-assessment as a survey will be delivered by Redcap survey, in person or remotely, or by telephone with researcher assistance. Completion of the survey will take approximately 10 minutes per week.
  Arms: Usual Care Control Group (UC)
Behavioral: Exit Interview — A semi-structured interview will be administered at 12 weeks to the intervention (EXE) group only to explore self-determination and efficacy, as well as intervention acceptability.
  Arms: Exercise Intervention Group (EXE)

SUMMARY:
The purpose of this study is to determine the effects of a multimodal exercise intervention on chemotherapy uptake in newly diagnosed pediatric, adolescent and young adult (AYA) Sarcoma patients.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of Sarcoma
2. Pediatric or AYA (12-39 years old)
3. Able to provide written informed consent
4. Able to speak, read, and understand English or Spanish
5. Initiating first-line systemic therapy (Doxorubicin, Ifosfamide, Gemcitabine, Docetaxel, Trabectedin, Vincristine, Irinotecan, Temozolomide, Topotecan, Etoposide, Dacarbazine, Pazopanib, Tazemetostat, Imatinib, Sunitinib, Pembrolizumab, Nivolumab, Ipilumumab, Regorafenib, Atezulimumab). Participants can be enrolled up to 90 days after starting firstline systemic therapy.
6. Approval from a medical oncology provider to participate.
7. Having not consistently (not equal to or more than 50% of the time) engaged in more than 90 minutes of moderate or 45 minutes of vigorous physical activity per week over the past 3 months
8. Having not consistently engaged in resistance training 2 or more days per week over the past 3 months

Exclusion Criteria:

1. < 12 or >39 years old
2. Unable to provide consent
3. Unable to read or understand English or Spanish
4. Oxygen-dependent
5. Unable to walk 2 blocks without assistance (excluding canes)
6. Unstable bone metastases
7. More than 90 days from initiation of first-line systemic therapy.
8. Presence of a severe medical condition or psychiatric condition or medications that would preclude participation of the study intervention, as determined by the patient's provider and study clinician.

Ages: 12 Years to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2027-09-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility of Participant Engagement at Time of Consent | Baseline
  Feasibility will be measured as the percentage of participants that consent and meet eligibility to participate between both the intervention and control arms. Criterion for success: At least (≥) 50% of all eligible participants consent to participate between both arms.
Feasibility of Participant Engagement at All Time Points | Up to 12 weeks
  Feasibility will be measured as the percentage of participants that adhere to and complete the arm-specific intervention and data collection at all time points between both the intervention and control arms. Criterion for success: Greater than (>) 70% of all eligible participants between both arms complete all scheduled assessments.
Acceptability of Participants that Feel Satisfied with Exercise Intervention | 12 weeks
  Acceptability will be measured as the percentage of participants that report satisfaction with the exercise intervention. Criterion for success: Greater than (>) 80% of all eligible participants complete the exercise intervention.

SECONDARY OUTCOMES:
Change in Chemotherapy RDI (Relative Dose Intensity) | Baseline, 12 weeks
  Change in chemotherapy relative dose intensity (RDI) at 12 weeks compared to baseline will be reported between both the intervention and control arms. RDI is the ratio of actual dose intensity to projected dose intensity, as a percentage or proportion of the amount of drug planned to deliver per weeks (mg/(m^2 x week)).

CONTACTS AND LOCATIONS:
Overall Officials: Tracy E Crane, PhD, RDN, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No